CLINICAL TRIAL: NCT01323556
Title: Mechanisms of CBT-Treatment Effects in Patients With Panic Disorder and Panic Disorder With Agoraphobia: The Role of Interoceptive Exposure
Brief Title: Mechanisms of Panic Disorders Treatment
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Prof. Dr. A. Hamm, University of Greifswald, Department of Clinical Psychology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AH 11.2009
Record Dates: First submitted 2011-03-03; First posted 2011-03-25 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-03

CONDITIONS: Panic Disorder; Agoraphobia; Panic Attacks
Keywords: Panic disorder; agoraphobia; panic attacks; exposure based learning; interoceptive exposure exercises; fear augmentation; in vivo exposure
MeSH Terms: conditions — Panic Disorder; Agoraphobia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exposure with fear augmentation (Experimental): exposure-based CBT, including interoceptive exposure and in-vivo exposure with fear augmentation by interoceptive exercises (e.g. hyperventilation)
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)
- Exposure without fear augmentation (Experimental): exposure-based CBT, including interoceptive and in-vivo exposure without fear augmentation during in-vivo exposure
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy (CBT) — 12 sessions of CBT including psychoeducation, behavioral analyses, interoceptive exposure and in-vivo exposure with interoceptive exposure during in vivo exposure
  Arms: Exposure with fear augmentation
Behavioral: Cognitive Behavioural Therapy (CBT) — 12 sessions of CBT including psychoeducation, behavioral analyses, interoceptive exposure and in-vivo exposure without additional fear augmenting strategies
  Arms: Exposure without fear augmentation

SUMMARY:
Investigation of mechanisms of exposure based learning by

1. Investigating the effects of fear augmentation by interoceptive exposure during in vivo exposure
2. Disentangling the effects of interoceptive exposure exercises in panic disorder

DETAILED DESCRIPTION:
The study aims on investigating the effect of fear augmentation during in-vivo exposure by adding interoceptive exposure (e.g., hyperventilation) in PD/AG patients. By comparing the fear augmentation group with the therapist-guided CBT exposure, and by measuring autonomic arousal during and between exposure sessions, it will be possible to study the mechanisms of exposure based learning. A second aim is to disentangle effects of specific interoceptive exposure exercises (e.g., respiratory vs. vestibular stimulation). Finally, by including patients without agoraphobic avoidance it will be possible to investigate whether interoceptive exposure alone will have any effect. This might open the door for early interventions for individuals after experiencing an initial panic attack to prevent the development of a severe panic disorder with agoraphobic avoidance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of panic disorder, panic disorder with agoraphobia OR initial panic attacks
* CGI ≥ 4 (except persons with initial panic attacks)
* Informed Consent

Exclusion Criteria:

* Acute suicidality
* Current substance use disorder
* Lifetime diagnosis of psychotic disorders, bipolar disorders, borderline personality disorders
* Severe medical condition (chronic conditions)
* Current psychotherapeutic or psychopharmacological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-10 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HARS) | up to 32 weeks (follow up)
  structured clinician rating assessing the severity of an anxiety disorder
Clinician Global Impression Scale (CGI) | up to 32 weeks (follow up)
  clinician rating assessing the severity of panic disorder and agoraphobia
Panic and Agoraphobia Scale (PAS) | up to 32 weeks (follow up)
  PAS is self-rating assessing panic disorder and agoraphobia severity with five factor analytic derived subscale scores (panic attacks, anticipatory anxiety, agoraphobic avoidance, health concerns, functional impairment) and a total score indicating the global severity. The questionnaire was specifically developed for monitoring changes during psychotherapy or psychopharmacological treatments.
Mobility Inventory | up to 32 weeks (follow up)
  Self-rating assessing the extent of situational avoidance. The questionnaire comprises 27 situations that have to be evaluated in regard to frequency of avoidance, when alone or when accompanied.
Number of panic attacks | up to 32 weeks (follow up)
  Number of panic attacks experienced during the last week is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Alfons O. Hamm, Prof. Dr., Principal Investigator — Institute for Psychology Ernst-Moritz-Arndt-University Greifswald Franz-Mehring-Str. 47; 17487 Greifswald, Germany; Thomas Lang, Dr., Study Director — Center for Clinical Psychology and Rehabilitation/ Christoph-Dornier-Foundation for Clinical Psychology University Bremen Grazer Str. 2b 28359 Bremen, Germany; Alexander L. Gerlach, Prof. Dr., Study Chair — Institute for Clinical Psychology and Psychotherapy WWU Münster Fliednerstr. 21 48149 Münster, Germany; Tilo Kirchner, Prof. Dr., Study Chair — Department of Psychiatry und Psychotherapy Philipps-University Marburg Rudolf-Bultmann- Straße 8 35039 Marburg, Germany; Georg W. Alpers, Prof. Dr., Study Chair — Institute for Biological Psychology, Clinical Psychology and Psychotherapy University Würzburg Marcusstrasse 9-11 97070 Würzburg, Germany
Locations (1):
- Prof. Dr. Alfons Hamm, Greifswald, Germany

REFERENCES:
- [Derived] Kunas SL, Hilbert K, Yang Y, Richter J, Hamm A, Wittmann A, Strohle A, Pfleiderer B, Herrmann MJ, Lang T, Lotze M, Deckert J, Arolt V, Wittchen HU, Straube B, Kircher T, Gerlach AL, Lueken U. The modulating impact of cigarette smoking on brain structure in panic disorder: a voxel-based morphometry study. Soc Cogn Affect Neurosci. 2020 Oct 8;15(8):849-859. doi: 10.1093/scan/nsaa103. PMID 32734299
- [Derived] Yang Y, Lueken U, Richter J, Hamm A, Wittmann A, Konrad C, Strohle A, Pfleiderer B, Herrmann MJ, Lang T, Lotze M, Deckert J, Arolt V, Wittchen HU, Straube B, Kircher T. Effect of CBT on Biased Semantic Network in Panic Disorder: A Multicenter fMRI Study Using Semantic Priming. Am J Psychiatry. 2020 Mar 1;177(3):254-264. doi: 10.1176/appi.ajp.2019.19020202. Epub 2019 Dec 16. PMID 31838872
- [Derived] Gechter J, Liebscher C, Geiger MJ, Wittmann A, Schlagenhauf F, Lueken U, Wittchen HU, Pfleiderer B, Arolt V, Kircher T, Straube B, Deckert J, Weber H, Herrmann MJ, Reif A, Domschke K, Strohle A. Association of NPSR1 gene variation and neural activity in patients with panic disorder and agoraphobia and healthy controls. Neuroimage Clin. 2019;24:102029. doi: 10.1016/j.nicl.2019.102029. Epub 2019 Oct 21. PMID 31734525
- [Derived] Forstner AJ, Awasthi S, Wolf C, Maron E, Erhardt A, Czamara D, Eriksson E, Lavebratt C, Allgulander C, Friedrich N, Becker J, Hecker J, Rambau S, Conrad R, Geiser F, McMahon FJ, Moebus S, Hess T, Buerfent BC, Hoffmann P, Herms S, Heilmann-Heimbach S, Kockum I, Olsson T, Alfredsson L, Weber H, Alpers GW, Arolt V, Fehm L, Fydrich T, Gerlach AL, Hamm A, Kircher T, Pane-Farre CA, Pauli P, Rief W, Strohle A, Plag J, Lang T, Wittchen HU, Mattheisen M, Meier S, Metspalu A, Domschke K, Reif A, Hovatta I, Lindefors N, Andersson E, Schalling M, Mbarek H, Milaneschi Y, de Geus EJC, Boomsma DI, Penninx BWJH, Thorgeirsson TE, Steinberg S, Stefansson K, Stefansson H, Muller-Myhsok B, Hansen TF, Borglum AD, Werge T, Mortensen PB, Nordentoft M, Hougaard DM, Hultman CM, Sullivan PF, Nothen MM, Woldbye DPD, Mors O, Binder EB, Ruck C, Ripke S, Deckert J, Schumacher J. Genome-wide association study of panic disorder reveals genetic overlap with neuroticism and depression. Mol Psychiatry. 2021 Aug;26(8):4179-4190. doi: 10.1038/s41380-019-0590-2. Epub 2019 Nov 11. PMID 31712720
- [Derived] Gottschalk MG, Richter J, Ziegler C, Schiele MA, Mann J, Geiger MJ, Schartner C, Homola GA, Alpers GW, Buchel C, Fehm L, Fydrich T, Gerlach AL, Gloster AT, Helbig-Lang S, Kalisch R, Kircher T, Lang T, Lonsdorf TB, Pane-Farre CA, Strohle A, Weber H, Zwanzger P, Arolt V, Romanos M, Wittchen HU, Hamm A, Pauli P, Reif A, Deckert J, Neufang S, Hofler M, Domschke K. Orexin in the anxiety spectrum: association of a HCRTR1 polymorphism with panic disorder/agoraphobia, CBT treatment response and fear-related intermediate phenotypes. Transl Psychiatry. 2019 Feb 4;9(1):75. doi: 10.1038/s41398-019-0415-8. PMID 30718541
- [Derived] Hommers LG, Richter J, Yang Y, Raab A, Baumann C, Lang K, Schiele MA, Weber H, Wittmann A, Wolf C, Alpers GW, Arolt V, Domschke K, Fehm L, Fydrich T, Gerlach A, Gloster AT, Hamm AO, Helbig-Lang S, Kircher T, Lang T, Pane-Farre CA, Pauli P, Pfleiderer B, Reif A, Romanos M, Straube B, Strohle A, Wittchen HU, Frantz S, Ertl G, Lohse MJ, Lueken U, Deckert J. A functional genetic variation of SLC6A2 repressor hsa-miR-579-3p upregulates sympathetic noradrenergic processes of fear and anxiety. Transl Psychiatry. 2018 Oct 19;8(1):226. doi: 10.1038/s41398-018-0278-4. PMID 30341278
- [Derived] Weck F, Grikscheit F, Hofling V, Kordt A, Hamm AO, Gerlach AL, Alpers GW, Arolt V, Kircher T, Pauli P, Rief W, Lang T. The role of treatment delivery factors in exposure-based cognitive behavioral therapy for panic disorder with agoraphobia. J Anxiety Disord. 2016 Aug;42:10-8. doi: 10.1016/j.janxdis.2016.05.007. Epub 2016 May 13. PMID 27235836
- [Derived] Hamm AO, Richter J, Pane-Farre C, Westphal D, Wittchen HU, Vossbeck-Elsebusch AN, Gerlach AL, Gloster AT, Strohle A, Lang T, Kircher T, Gerdes AB, Alpers GW, Reif A, Deckert J. Panic disorder with agoraphobia from a behavioral neuroscience perspective: Applying the research principles formulated by the Research Domain Criteria (RDoC) initiative. Psychophysiology. 2016 Mar;53(3):312-22. doi: 10.1111/psyp.12553. PMID 26877119
- See also: Related Info — http://www.paniknetz.de/